CLINICAL TRIAL: NCT00093249
Title: Efficacy Study of Clevidipine Assessing Its Preoperative Antihypertensive Effect in Cardiac Surgery (ESCAPE-1)
Brief Title: Study of Clevidipine Assessing Its Preoperative Antihypertensive Effect in Cardiac Surgery (ESCAPE-1)
Acronym: ESCAPE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMC-CLV-03-01; ESCAPE-1 (Other: Sponsor)
Record Dates: First submitted 2004-10-05; First posted 2004-10-07 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: Pre-operative hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clevidipine (Experimental): Clevidipine was administered in a blinded fashion by intravenous (IV) infusion, starting at a rate of 0.4 μg/kg/min (non weight-based equivalent is 2 mg/hr) and titrating upward, as tolerated, in doubling increments approximately every 90 seconds to achieve the desired blood pressure-lowering effect. Up-titration to 3.2 μg/kg/min (16 mg/hr) was allowed. Infusion rates above 3.2 μg/kg/min could be used, guided by the patient's response, by increasing in serial increments of 1.5 μg/kg/min up to the maximum recommended clevidipine infusion rate of 8.0 μg/kg/min. Clevidipine was to be administered for a minimum of 30 minutes, unless bailout occurred, and up to a maximum of one hour.
  Interventions: Drug: clevidipine
- placebo (Placebo Comparator): Placebo consisted of 20% lipid emulsion (the same lipid vehicle used for clevidipine) administered in a blinded fashion intravenously following the same study drug administration guidelines as with clevidipine study drug administration guidelines. As with clevidipine, placebo was to be administered for a minimum of 30 minutes, unless bailout occurred, and up to a maximum of one hour.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clevidipine — Clevidipine (0.5 mg/mL in 20% lipid emulsion)will be administered intravenously at an initial infusion rate of 0.4 µg/kg/min and will be titrated, as tolerated, at the discretion of the investigator, in doubling increments approximately every 90 seconds up to a maximum of 3.2 µg/kg/min, in order to achieve the desired blood pressure lowering effect. Clevidipine may be titrated upwards or downwards and may be temporarily interrupted and restarted to attain the desired blood pressure effect. The maximum study drug infusion rate of 8.0 µg/kg/min may not be exceeded.
  Other Names: clevidipine, Cleviprex
  Arms: clevidipine
Drug: placebo — Placebo (20% lipid emulsion - vehicle) will be administered intravenously in a fashion identical to clevidipine as described above.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the efficacy of clevidipine injection versus placebo in treating preoperative hypertension.

DETAILED DESCRIPTION:
Initiation of study drug infusion will commence with the occurrence of protocol-defined preoperative hypertension (SBP > 160 mmHg) as measured via an indwelling arterial line.

The study drug (clevidipine or placebo) may be administered to treat hypertension until one hour has elapsed, or until induction of anesthesia, whichever occurs first.

The primary endpoint of bailout described (as defined per protocol) as bailout for lack of efficacy, bailout for safety reason or bailout due to treatment failure will be determined during the 30-minute period from study drug initiation.

ELIGIBILITY:
Pre-randomization Inclusion Criteria:

* Provide written informed consent before initiation of any study-related procedures.
* Be at least 18 years of age
* Be scheduled for cardiac surgery (including Coronary Artery Bypass Grafting [CABG], Off Pump Coronary Artery Bypass [OPCAB], Minimally Invasive Direct Coronary Artery Bypass [MIDCAB] surgery, and/or valve replacement/repair procedures)
* Have a recent history (within 6 months of randomization) of hypertension requiring treatment with antihypertensive medication(s) or be actively hypertensive upon admission

Pre-randomization Exclusion Criteria:

* Women of child-bearing potential (unless they have a negative pregnancy test)
* Recent cerebrovascular accident (within 3 months before randomization)
* Known intolerance to calcium channel blockers
* Allergy to soybean oil or egg lecithin (components of the lipid vehicle)
* Pre-existing left bundle branch block or permanent ventricular pacing
* Any other disease or condition, which, in the judgment of the investigator would place a patient at undue risk by being enrolled in the trial.
* Participation in another therapeutic drug or therapeutic device trial within 30 days of starting study

Post-randomization Inclusion Criteria:

* After the insertion of an arterial line, the patient is determined to meet the per protocol preoperative definition of hypertension, i.e. systolic blood pressure (SBP) > 160 mmHg
* It is the investigator's intent to lower the patient's SBP by a minimum of 15% from its baseline value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-01; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Incidence of bailout during 30-minute treatment period | During the first 30 minutes post study drug initiation
  discontinuation of study drug categorized according to the following reasons:
  * Bailout for lack of efficacy
  * Bailout for safety reason(s)
  * Bailout due to treatment failure

SECONDARY OUTCOMES:
Median time to target SBP lowering effect (defined as a reduction by 15% or more) | During the first 30 minutes post study drug initiation
Mean arterial pressure (MAP) change from baseline | During the first 30 minutes post study drug initiation
Heart rate change from baseline | During the first 30 minutes post study drug initiation
Incidence of bailout by causality | During the first 30 minutes post study drug initiation

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Cardio-Thoracic Surgeons, PC, Birmingham, Alabama
  - St Vincent Medical Center, Los Angeles, California
  - Discovery Alliance - Hudson, Hudson, Florida
  - Discovery Alliance - Sacred Heart Hospital, Pensacola, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - MacNeal Hospital, Berwyn, Illinois
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Christ Hospital, The Linder Clinical Trial Center, Cincinnati, Ohio
  - Memorial Herman Memorial City Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - Houston Northwest Medical Center, Houston, Texas
  - Swedish Hospital Medical Center, Seattle, Washington

REFERENCES:
- [Result] Levy JH, Mancao MY, Gitter R, Kereiakes DJ, Grigore AM, Aronson S, Newman MF. Clevidipine effectively and rapidly controls blood pressure preoperatively in cardiac surgery patients: the results of the randomized, placebo-controlled efficacy study of clevidipine assessing its preoperative antihypertensive effect in cardiac surgery-1. Anesth Analg. 2007 Oct;105(4):918-25, table of contents. doi: 10.1213/01.ane.0000281443.13712.b9. PMID 17898366